CLINICAL TRIAL: NCT06031129
Title: Effectiveness of Butorphanol in Alleviating Postoperative Visceral Pain Following Microwave Ablation for Hepatic Tumor: A Multicentral, Randomized, Placebo-Controlled Trial
Brief Title: Butorphanol in Pain Following Ablation for Hepatic Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bibo Wang (Other)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Sponsor-Investigator, Bibo Wang, Principal Investigator of Oncology Department, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Jinling WBB
Record Dates: First submitted 2023-08-29; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Visceral Pain; Microwave Ablation; Hepatic Tumor
MeSH Terms: conditions — Visceral Pain; Carcinoma, Hepatocellular | interventions — Butorphanol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Butorphanol (Experimental)
  Interventions: Drug: Butorphanol
- normal saline (Placebo Comparator)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Butorphanol — The pharmacological attributes of Butorphanol, characterized by its mild impact on cardiopulmonary dynamics and demonstrated efficacy in attenuating mechanical traction-induced discomfort, culminate in an ameliorative effect on postoperative nausea and vomiting rates. Importantly, it substantively attenuates visceral postoperative pain. However, sedation can also cause dizziness, drowsiness, and other adverse reactions during recovery
  Arms: Butorphanol
Drug: normal saline — normal saline contain 0.9% NaCl sodium.
  Arms: normal saline

SUMMARY:
The objective of this investigation was to evaluate the influence of Butorphanol on postoperative pain mitigation in patients undergoing microwave ablation for hepatic tumor. Employing a rigorously designed multicentral, randomized, and placebo-controlled format, patients subjected to microwave ablation were assigned randomly to either Butorphanol (experimental group) or normal saline (control group). Primary outcomes encompassed intraoperative pain levels assessed through patient-driven evaluation utilizing a 10-point visual analog scale (VAS). Secondary outcomes included postoperative pain levels at the 6-hour mark (VAS) and comprehensive pain assessment outcomes.

ELIGIBILITY:
Inclusion Criteria:

patients performing Microwave Ablation sign the informed consent

Exclusion Criteria:

Patients with a body mass index > 30 kg/m2 a history of depression opioid dependence poorly controlled hypertension (systolic blood pressure > 180 mmHg) myocardial infarction severe liver disease significant abdominal pain before surgery patients with sensory system or language dysfunctions who could not cooperate to complete the scale pregnant women.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Visceral Pain | during the surgery
  VAS score of visceral pain

SECONDARY OUTCOMES:
Visceral Pain | 6-hour after surgery
  VAS score of visceral pain

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hosipiatl, Nanjing, Jiangsu, China